CLINICAL TRIAL: NCT05142787
Title: A Prospective, Multi Center, International, Open Label Study of the Use of Magseed Pro(R) Markers and Sentimag(R) Gen3 to Localize Breast Lesions and Suspicious/biopsy-proven Positive Lymph Nodes in Breast Cancer Patients
Brief Title: Magseed Pro(R)/ Sentimag(R) Gen3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endomagnetics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EU001
Record Dates: First submitted 2021-11-08; First posted 2021-12-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
Keywords: Magseed Pro; Sentimag Gen3
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- axillary lymph nodes requiring localisation prior to surgical excision (Other): The Magseed Pro® marker is intended to be placed percutaneously in suspicious/biopsy proven positive axillary lymph nodes under imaging guidance to mark tissue intended for selective surgical removal.
  The Magseed Pro® marker is localised using the Sentimag® Gen3 system handheld probes and surgically removed within/from the target tissue.
  Interventions: Device: Magseed Pro(R) and Sentimag(R) Gen3 by Endomagnetics
- breast lesions requiring localisation (Other): The Magseed Pro® marker is intended to be placed percutaneously in breast lesions under imaging guidance to mark tissue intended for selective surgical removal.
  The Magseed Pro® marker is localised using the Sentimag® Gen3 system handheld probes and surgically removed within/from the target tissue.
  Interventions: Device: Magseed Pro(R) and Sentimag(R) Gen3 by Endomagnetics

INTERVENTIONS:
Device: Magseed Pro(R) and Sentimag(R) Gen3 by Endomagnetics — placement of Magseed Pro & localisation with Sentimag Gen3 in axillary lymph nodes and/or breast lesions

SUMMARY:
The purpose of this study is to provide prospective evidence that the Magseed Pro® marker /Sentimag® Gen3 system is safe and effective for marking A. suspicious/biopsy-proven positive axillary lymph nodes; and B. soft tissue lesions including cancer and pre-cancerous change in the breast

DETAILED DESCRIPTION:
The purpose of this study is to provide prospective evidence that the Magseed Pro® marker /Sentimag® Gen3 system is safe and effective for marking A. suspicious/biopsy-proven positive axillary lymph nodes; and B. soft tissue lesions including cancer and pre-cancerous change in the breast The devices used in this clinical trial are the Magseed Pro® marker and Sentimag® Gen3 system by Endomagnetics Limited.

The Endomag Magseed Pro® Marker System is intended to be placed within the target soft tissue prior to planned surgical removal. The marker, when used in conjunction with the Sentimag® Gen 3 System, can be used as a guide for the surgeon to follow in the excision of tissue. The Sentimag® Gen3 Magnetic Localisation System when used with the Magseed family of markers is indicated to assist in localising soft tissue lesions.

The study design is a multicentre international prospective, open label, study of Magseed Pro® marker and Sentimag® Gen3 system in patients with breast and/or lymph node pathology with:

A. axillary lymph nodes requiring localisation prior to surgical excision (suspicious and/or biopsy proven lymph node or other pathology indicating removal) and/or B. breast lesions requiring localisation

Patients will have the Magseed Pro® marker placed to mark A. surgical excision of suspicious/biopsy-proven axillary lymph node as part of a targeted lymph node biopsy procedure AND/OR B. breast lesions in patients undergoing surgical excision of the targeted breast lesion The Magseed Pro® marker will be localised using the Sentimag® Gen3 system and therafter surgically removed with the target tissue.

This study will enrol 224 patients; 112 with Magseed Pro® marker placed to mark breast lesions and 112 with Magseed Pro® marker placed to mark nodes.

The expected duration of enrolment is approximately 9 months across all sites with each individual subject's participation lasting approximately 1-38 weeks after enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Participant is aged 18 years or older at the time of consent.
* Patients requiring breast lesion/axillary node marking and excision

Exclusion Criteria:• Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period. A pregnancy test is required for all women of childbearing potential within 7 days before enrolment.

* Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical trial or to comply with follow up requirements, or impact the scientific soundness of the clinical trial results
* Known hypersensitivity to Nitinol
* Subject has current active infection at the implantation site in the breast (per investigator discretion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The primary endpoints are the retrieval rates of the Magseed Pro® marker with the target lesion within the initial excised specimen for A.) axillary lymph nodes B.) breast lesions A.) axillary lymph nodes. B.) breast lesions | time of surgery
  This is defined as the number of patients with successful Magseed Pro® marker placement as demonstrated on imaging, in whom the Magseed Pro® marker and the associated lymph node and/ or lesion is retrieved, divided by the total number of subjects.

SECONDARY OUTCOMES:
Tissue response (unexpected and expected) | time of surgery
  EXPECTED Early (up to 2 days) - acute inflammation in the form of neutrophils with lymphocytes and some associated haemorrhage.
  Late (>2 days) - active chronic inflammation in the form of neutrophils, lymphocytes, macrophages together with a fibroblastic response. Likely a foreign body reaction with increased numbers of histiocytes and some multinucleated giant cells. Possible granuloma formation (foreign body type). Scattered eosinophils. Later scarring (after 1-2 weeks) with fibrosis. Possible fat necrosis.
  UNEXPECTED Early and Late -
  • Very florid fibroblastic response with granulation tissue formation that mimics malignancy (nodular fasciitis-like), which may need immunohistochemical tests to differentiate between reactive chan
Presence of unexpected histological tissue response for short- and long-term use of Magseed Pro marker | time of surgery
  UNEXPECTED HISTOLOGICAL RESPONSE Early and Late -
  • Very florid fibroblastic response with granulation tissue formation that mimics malignancy (nodular fasciitis-like), which may need immunohistochemical tests to differentiate between reactive chan
Rate of device-related AE's and SAE's | through study completion, an average of 38 weeks
  Rate of device-related AE's and SAE's
Retrieval rate for all lesions | time of surgery
  Retrieval rate for all lesions (including target, non-target lesions and multiple lesions per patient) out of the total number of lesions with a Magseed Pro® marker placement. Non-target lesions include additional marked lesions which weren't defined as the target for the primary endpoint and any marked lesions from patients undergoing long term node retrieval.
Retrieval rate for all nodes | time of surgery
  Retrieval rate for all nodes (including multiple nodes per patient where applicable) out of the total number of nodes with a Magseed Pro® marker placement.
Per lesion retrieval rate for target excised specimens | time of surgery
  Per lesion retrieval rate for target excised specimens
Per lesion retrieval rate for all excised specimens | time of surgery
  Per lesion retrieval rate for all excised specimens
Per lesion retrieval rate for all lesion | time of surgery
  Per lesion retrieval rate for all lesion
Per lesion retrieval rate for all nodes | time of surgery
  Per lesion retrieval rate for all nodes
Per patient retrieval rate for Magseed Pro® marker placed prior to neo-adjuvant therapy and retrieved post neo-adjuvant therapy | time of surgery
  Per patient retrieval rate for Magseed Pro® marker placed prior to neo-adjuvant therapy and retrieved post neo-adjuvant therapy
Per lesion retrieval rate for Magseed Pro® marker placed prior to neo-adjuvant therapy and retrieved post neo-adjuvant therapy. | time of surgery
  Per lesion retrieval rate for Magseed Pro® marker placed prior to neo-adjuvant therapy and retrieved post neo-adjuvant therapy.
Per patient retrieval rate for Magseed Pro® marker where retrieval surgery is within 30 days of placement. | time of surgery
  Per patient retrieval rate for Magseed Pro® marker where retrieval surgery is within 30 days of placement.
Per lesion retrieval rate for Magseed Pro® marker where retrieval surgery is within 30 days of placement. | time of surgery
  Per lesion retrieval rate for Magseed Pro® marker where retrieval surgery is within 30 days of placement.
Per patient retrieval rate for Magseed Pro® marker where retrieval surgery is greater than 30 days after placement | time of surgery
  Per patient retrieval rate for Magseed Pro® marker where retrieval surgery is greater than 30 days after placement
Per lesion retrieval rate for Magseed Pro® marker where retrieval surgery is greater than 30 days after placement. | time of surgery
  Per lesion retrieval rate for Magseed Pro® marker where retrieval surgery is greater than 30 days after placement.
Per lesion retrieval rate for target excised specimens (i.e., lesions plus nodes) where Magtrace® Tracer is present in the target node or in the region of the target lesion. | time of surgery
  Per lesion retrieval rate for target excised specimens (i.e., lesions plus nodes) where Magtrace® Tracer is present in the target node or in the region of the target lesion.
Per lesion retrieval rate for all excised specimens (i.e., lesions plus nodes) where Magtrace® Tracer is present in the target node or in the region of the target lesion. | time of surgery
  Per lesion retrieval rate for all excised specimens (i.e., lesions plus nodes) where Magtrace® Tracer is present in the target node or in the region of the target lesion.
Per lesion retrieval rate for target lesions where Magtrace® Tracer is present in the region of the target lesion. | time of surgery
  Per lesion retrieval rate for target lesions where Magtrace® Tracer is present in the region of the target lesion.
Per lesion retrieval rate for all lesions where Magtrace® Tracer is present in the region of the lesion. | time of surgery
  Per lesion retrieval rate for all lesions where Magtrace® Tracer is present in the region of the lesion.
Per node retrieval rate for target nodes where Magtrace® Tracer is present in the target node. | time of surgery
  Per node retrieval rate for target nodes where Magtrace® Tracer is present in the target node.
Per node retrieval rate for all nodes where Magtrace® Tracer is present in the node. | time of surgery
  er node retrieval rate for all nodes where Magtrace® Tracer is present in the node.
Interventionist rated ease of Magseed Pro® marker placement by the interventionist | seed placement
  5 point Likert scale, very easy = 5, very difficult = 1
Rate of deployment failure | seed placement
  A Magseed Pro is not deployed from the needle, or is accidentally deployed prior to use in the patient
  • Success rate of seed placement:
  * Accurate: Within the breast lesion or clipped lymph node. For lesions less than 5 mm in size the marker may not necessarily be within the excised specimen but should be within 10mm1 of the lesion.
  * Inadequate: Not in the targeted lesion or clipped lymph node determined by placement imaging requiring additional marker placement
Surgeon rated ease of intra-operative localisation | time of surgery
  5 point Likert scalevery easy = 5, very difficult = 1
Magtrace® Tracer counts for excised lymph nodes during SLNB procedures | time of surgery
  Magtrace® Tracer counts for excised lymph nodes during SLNB procedures
Re-excision rate (i.e., second procedure required). With reason for second procedure. | time of surgery
  Re-excision rate (i.e., second procedure required). With reason for second procedure.
Success rate of maintained marker position at the time of removal as determined by specimen X-ray and or Sentimag Gen3 system. | time of surgery
  * Accurate: Magseed Pro® marker within the target lesion or marked lymph node.
  * Inadequate: Magseed Pro® marker not within the target lesion or marked lymph node

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Paepke, Dr, Principal Investigator — The technical university of Munich
Locations (6):
- Germany (3):
  - Marienhospital Bottrop GmbH, Bottrop
  - AGAPLESION Markus Frankfurter Diakonie Kliniken gGmbH, Frankfurt
  - Technical University Munich, Munich
- United Kingdom (3):
  - Guy's Hospital, London
  - Royal Marsden Hospital, London
  - University Hospital South Manchester, Manchester

IPD SHARING:
Plan to Share IPD: No